CLINICAL TRIAL: NCT05360784
Title: The Efficacy and Safety of Brimonidine Tartrate Ophthalmic Solution 0.025% Preservative-Free Formulation With Lumify® 0.025% in Adult Subjects With Ocular Redness
Brief Title: "Efficacy and Safety of Brimonidine Tartrate Preservative-Free Formulation in Adults With Ocular Redness"
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 908
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Results first posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2023-06

CONDITIONS: Ocular Redness
MeSH Terms: interventions — Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brimonidine tartrate preservation-free (Experimental): Brimonidine tartrate ophthalmic solution 0.025% preservative-free formulation
  Interventions: Drug: Brimonidine tartrate ophthalmic solution 0.025% preservative-free formulation
- Lumify® (Active Comparator): Lumify® (brimonidine tartrate ophthalmic solution 0.025%)
  Interventions: Drug: Lumify® (brimonidine tartrate ophthalmic solution 0.025%)

INTERVENTIONS:
Drug: Brimonidine tartrate ophthalmic solution 0.025% preservative-free formulation — Brimonidine tartrate ophthalmic solution 0.025% preservative-free formulation. Participants will instill 1 drop of the assigned investigational drug in each eye 4 times a day approximately 4 hours apart for up to 4 consecutive weeks.
  Arms: Brimonidine tartrate preservation-free
Drug: Lumify® (brimonidine tartrate ophthalmic solution 0.025%) — Lumify® (brimonidine tartrate ophthalmic solution 0.025%). Participants will instill 1 drop of the assigned investigational drug in each eye 4 times a day approximately 4 hours apart for up to 4 consecutive weeks.
  Arms: Lumify®

SUMMARY:
This is a multi-center, double-masked, randomized, active-controlled, parallel-group, efficacy and safety study that will enroll 386 participants at up to six clinical sites. Participants with ocular redness will be randomized to receive either brimonidine tartrate ophthalmic solution 0.025%, preservative-free formulation, or Lumify® (brimonidine tartrate ophthalmic solution 0.025%). Participants will be treated with study drug for approximately 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age at the time of Informed Consent signing of either gender and any race or ethnicity;
2. Provide written informed consent and sign the HIPAA form;
3. Be willing and able to follow all instructions and attend all study visits;
4. Have a history of vasoconstrictor (redness relief drops) use within the last 6 months, or a desire to use OTC vasoconstrictors for redness relief;
5. Be able to self-administer eye drops satisfactorily or have a subject's care provider at home1 routinely available for this purpose;
6. (If female and of childbearing potential) agree to have urine pregnancy testing performed at Visit 1 (must be negative) and at exit visit; must not be lactating; and must agree to use at least 1 medically acceptable form of birth control2 throughout the study duration and for at least 14 days prior to the first dose of study drug (Visit 1) and for 1 month after the last dose of investigational drug. Note: Women considered capable of becoming pregnant include all females who have experienced menarche and have not experienced menopause (as defined by amenorrhea for greater than 12 consecutive months) and have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy);
7. (If male and with female partner of childbearing potential) must use at least 1 medically acceptable form of birth control3;
8. A calculated best-corrected (if necessary) visual acuity of 0.3 logMAR or better in each eye, as measured using an ETDRS chart;
9. At Visit 1 (Baseline), show a baseline redness score >1 unit (ie, greater than 1 unit) in both eyes on a 0 to 4 unit scale as scored by the Investigator using the Investigator Ocular Redness Scale;
10. Have stable ocular health (defined as no ocular conditions requiring therapy or surgical intervention during the study).

Exclusion Criteria:

1. Have known contraindications or sensitivity to the use of any of the investigational drug(s) or their components, or any other medications required by the protocol;
2. Have had ocular surgical intervention within 3 months prior to screening or during the study and/or a history of refractive surgery within the past 6 months;
3. Have the presence of an active ocular infection (bacterial, viral, or fungal) or positive history of an ocular herpetic infection at any visit;
4. Use any of the following disallowed medications during the period indicated prior to screening and for the duration of the study:

   * All topical ophthalmic agents including artificial tear products, eye whiteners (e.g., vasoconstrictors), ocular decongestants, ocular antihistamines, ocular corticosteroids, dilating drops, (excluding dilated ophthalmoscopy exam at Visit 1) and contact lenses: 5 days
   * Systemic antihistamines or decongestants: 7 days
   * Systemic corticosteroids or cancer chemotherapy, and/or any other systemic medications which the investigator feels may confound study data, or interfere with subject's study participation: 14 days
5. Have prior (within 7 days of beginning investigational drug) or currently active significant illness that could compromise participation, in the opinion of the investigator;
6. Have prior (within 30 days of beginning investigational drug) or anticipated concurrent use of an investigational drug or device during the study period;
7. Have an ocular or systemic condition or a situation which, in the investigator's opinion, may put the subject at increased risk, confound study data, or interfere significantly with the subject's study participation;
8. Have planned surgery (ocular or systemic) during the trial period or within 30 days after the study period;
9. Be currently breast feeding or planning to breast feed during the study period or is a female who is currently pregnant, is planning a pregnancy, or has a positive urine pregnancy test at Visit 1;
10. Have a diagnosis of ocular hypertension or glaucoma at screening;
11. Have symptoms that, in the opinion of the investigator, may be associated with COVID-19 or in the last 14 days came into contact with someone diagnosed with COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Donatello, Study Director — Bausch & Lomb Incorporated
Locations (6):
- United States (6):
  - Bausch Site 04, Colorado Springs, Colorado
  - Bausch Site 05, Louisville, Kentucky
  - Bausch Site 01, Andover, Massachusetts
  - Bausch Site 03, Shelby, North Carolina
  - Bausch Site 02, Memphis, Tennessee
  - Bausch Site 06, Clinton, Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Toyos M, DiVito M, Messmer EM, McGee S, Peterson J, Patel A, Pattar G, Evans DG, Vollmer PM, Wesley G. A Multicenter Randomized Double-Masked Study Comparing Preservative-free Brimonidine Tartrate Ophthalmic Solution 0.025% with LUMIFY(R) 0.025% for Ocular Redness in Adults. Ophthalmol Ther. 2025 Sep;14(9):2283-2299. doi: 10.1007/s40123-025-01194-z. Epub 2025 Jul 25. PMID 40711722

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brimonidine Tartrate Preservation-free | Lumify®
Started | 190 | 190
Completed | 165 | 179
Not Completed | 25 | 11
Not completed — Discontinued | 25 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brimonidine Tartrate Preservation-free | Lumify® | Total
Number analyzed (Participants) | 190 | 190 | 380
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 114 | 106 | 220
  >=65 years | 76 | 84 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (14.65) | 59.5 (14.76) | 59 (14.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 125 | 267
  Male | 48 | 65 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 17 | 29
  Not Hispanic or Latino | 178 | 173 | 351
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 5
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 46 | 43 | 89
  White | 138 | 138 | 276
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 190 | 190 | 380

OUTCOME MEASURES:

1. Primary Outcome: Ocular Redness
Description: Ocular redness score evaluated by the investigator from 5 minutes to 240 minutes after investigational drug instillation (0-4 unit scale, where 0 = None and 4 = Extremely severe).
Time Frame: Assessed at 5, 15, 30, 60, 90,120,180, 240 minutes post instillation.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Brimonidine Tartrate Preservation-free | Lumify®
Number analyzed (Participants) | 190 | 190
score on a scale
  5 minutes Post Instillation | 0.46 (0.039) | 0.53 (0.041)
  15 minutes Post Instillation | 0.40 (0.038) | 0.49 (0.041)
  30 minutes Post Instillation | 0.42 (0.038) | 0.50 (0.041)
  60 minutes Post Instillation | 0.47 (0.040) | 0.52 (0.041)
  90 minutes Post Instillation | 0.54 (0.043) | 0.58 (0.044)
  120 minutes Post Instillation | 0.64 (0.046) | 0.67 (0.046)
  180 minutes Post Instillation | 0.79 (0.046) | 0.84 (0.049)
  240 minutes Post Instillation | 0.99 (0.047) | 0.98 (0.049)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 36 days.
Arm/Group | Brimonidine Tartrate Preservation-free | Lumify®
All-Cause Mortality (participants affected / at risk) | 0/188 | 0/190
Serious Adverse Events (participants affected / at risk) | 0/188 | 1/190
Other Adverse Events (participants affected / at risk) | 13/188 | 18/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brimonidine Tartrate Preservation-free (N=188) | Lumify® (N=190)
Sepsis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brimonidine Tartrate Preservation-free (N=188) | Lumify® (N=190)
Visual acuity reduced (Eye disorders) | 0 | 4
Covid 19 (Infections and infestations) | 5 | 2
Sinusitis (Infections and infestations) | 2 | 6
Instillation site pain (General disorders) | 6 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact Sponsor directly for details

DOCUMENTS (2):
  • Study Protocol (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT05360784/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-16): https://cdn.clinicaltrials.gov/large-docs/84/NCT05360784/SAP_001.pdf